CLINICAL TRIAL: NCT01573247
Title: A Phase 1/2, Open-Label, Multi-Center Dose Escalation, Safety and Tolerability Study of AKN-028 in Patients With Acute Myelogenous Leukemia (AML)
Brief Title: Safety Study of AKN-028 in Patients With Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: During the study two patients have experienced serious liver events related to AKN-028. The risk-benefit balance was judged to be negative.
Sponsor: Akinion Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKN001; 2011-003285-33 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-09 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Refractory Acute myeloid leukemia; FLT3 inhibitor; kinase inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-3-(1H-indol-5-yl)-5-pyridin-4-yl-pyrazine-2,3-diamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AKN-028 (Experimental)
  Interventions: Drug: AKN-028

INTERVENTIONS:
Drug: AKN-028 — Part 1 of the study is a sequential dose-escalation evaluation of AKN-028. Part 1 started as an accelerated intra-patient dose escalation design in one patient at a time (the N=1 portion), and has switched to standard 3 + 3 design with inter-cohort dose escalation when AUC of 12 μM*hrs has been reached. Starting dose of AKN-028 was 60 mg twice a day.
  During Part 2 of the study AKN-028 will be administered at the dose level selected in Part 1. Patients will be treated for a maximum of 3 cycles (first cycle of 14 days followed by 2 cycles of 21 days), with at least a 7-day treatment-free period between cycles. Patients with significant benefit after 3rd cycle may continue treatment at discretion of the investigator for as long as the patient continues to show significant benefit.

SUMMARY:
This Phase 1/2 study consists of two parts. The purpose of Part 1 of the study is to examine the safety and tolerability of AKN-028 and to determine the recommended dose of AKN-028 for further evaluation in Part 2 of the study in patients with Acute Myelogenous Leukemia (AML). The purpose of Part 2 of the study is to determine safety and efficacy in patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to Screening;
* Male or female patients, age ≥ 18 years;
* For females of childbearing potential, a negative urine pregnancy test must be obtained
* Confirmed diagnosis of AML (≥ 20% blasts in bone marrow and / or peripheral blood) according to World Health Organization (WHO) classification [2] and meeting at least one of the following:

  1. Newly diagnosed AML, but according to the clinical judgment of the principal investigator, patient is not a candidate for induction chemotherapy because of age, comorbidity, performance status, or other factors;
  2. AML in first relapse with WBC < 60,000/mm3 and ineligible for further intensive induction chemotherapy;
  3. AML in second relapse with low peripheral blast count (< 10,000/mm3) and with WBC < 60,000/mm3 and ineligible for intensive induction chemotherapy;
  4. Primary refractory disease, here defined as patients with AML not having achieved CR following up to 2 courses of chemotherapy for enrollment in Part 1 and patients with AML refractory following 1 course of chemotherapy for enrollment in Part 2;

Note: Severe neutropenia per se (up to Grade 4) should be accepted if it is likely to be related to the AML. However, the severe neutropenia may be due to the recently administered chemotherapy (e.g. cytarabin). It may be prudent to perform a new bone marrow examination. In case the marrow is hypoplastic (due to cytarabin) the screening should be postponed and G-CSF should be administered for a short period and then the patient should be re-evaluated. In case the bone marrow is not hypoplastic but rather infiltrated with AML cells the patient can be screened.

* Performance status of 0-3 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale;
* Adequate organ function, including the following:

  * Serum creatinine ≤ 2.0 mg/dL (176.8 mMol/L) during screening;
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x the upper limits of normal (ULN) during screening; and
  * Total bilirubin ≤1.5 x ULN during screening.

Exclusion Criteria:

* Patients who are candidates for induction chemotherapy for AML
* Total WBC count ≥ 60,000/mm3;
* Evidence of active central nervous system (CNS) leukemia;
* Evidence of blast-phase chronic myelogenous leukemia (CML);
* Histological or cytogenetic diagnosis of AML with M3 subtype (Acute Promyelocytic Leukemia);
* Lack of recovery of non-hematological toxicity from systemic therapy for the underlying hematologic condition;
* Previous or concurrent malignancy except non-invasive non-melanoma skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 2 years prior to study entry; this exclusion does not refer to the disease (AML) under study;
* Uncontrolled systemic infection (viral, bacterial, or fungal);
* Uncontrolled disseminated intravascular coagulation;
* Known positive serology for human immunodeficiency virus;
* Clinically significant cardiac dysfunction (New York Heart Association Class 3 or 4) at the time of screening, or a history of myocardial infarction or heart failure within 3 months preceding the first dose of AKN-028;
* Chronic Graft versus Host Disease (GVHD) with the exception of mild (Grade 1) skin or oral GVHD;
* Major surgery within the 28 days preceding the first dose of AKN-028;
* Concomitant administration of any other anti-leukemia or anti-neoplastic therapy (during the screening period, hydroxyurea is allowed for ≤ 7 days before Cycle 1, as well as for ≤ 7 days between cycles);
* Concomitant treatment with immunotherapy, or any investigational agent within 28 days preceding the first dose of AKN-028, or lack of recovery from toxicity of such treatment;
* Active autoimmune disease requiring immunosuppressive therapy;
* Radiotherapy, or lack of recovery of any radiotherapy-related acute toxicity, within the 28 days preceding the first dose of AKN-028;
* Previous treatment in any clinical study with AKN-028, any other FLT-3 inhibitor, or any other c-Kit inhibitor;
* Female patients who are pregnant or breast-feeding;
* Male, or female patients of childbearing potential, unwilling to use an approved, effective means of contraception (e.g., oral contraception, barrier contraception, intrauterine device) in accordance with the investigator's standards;
* Known current drug or alcohol abuse;
* Active viral Hepatitis B and /or C;
* Other severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that, in the opinion of the investigator, may compromise the safety of the patient during the study, affect the patient's ability to complete the study, or interfere with interpretation of study results;
* Any condition, which is judged by the Investigator to be inappropriate for study participation, including an inability to communicate or cooperate with the Investigator and the requirements of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic profiles | up to 3 months
Adverse Events | up to 3 months
  Safety follow up

SECONDARY OUTCOMES:
Response | participants will be followed for the duration of up to 3 months
  Biological respons

CONTACTS AND LOCATIONS:
Overall Officials: Martin Höglund, MD, PhD, Principal Investigator — Dept of Hematology, Uppsala University Hospital
Locations (8):
- Czechia (2):
  - University Hospital Brno, Brno
  - University Hospital Kralovske Vinohrady, Prague
- Poland (2):
  - MTZ Clinical Research Inc., Warsaw
  - Institute of Hematology and Transfusion Medicine, Warsaw
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Orebro University Hospital, Örebro
  - Uppsala University Hospital, Uppsala
- St.Bartholomew's Hospital, West Smithfield, United Kingdom

REFERENCES:
- [Derived] Eriksson A, Kalushkova A, Jarvius M, Hilhorst R, Rickardson L, Kultima HG, de Wijn R, Hovestad L, Fryknas M, Oberg F, Larsson R, Parrow V, Hoglund M. AKN-028 induces cell cycle arrest, downregulation of Myc associated genes and dose dependent reduction of tyrosine kinase activity in acute myeloid leukemia. Biochem Pharmacol. 2014 Jan 15;87(2):284-91. doi: 10.1016/j.bcp.2013.10.022. Epub 2013 Nov 4. PMID 24200998